CLINICAL TRIAL: NCT04204460
Title: Electromyographic Evaluation of Quadriceps During Eccentric Decline Squat: An Investigation of the Effect of Decline Angle and Arc of Motion
Brief Title: Electromyographic Evaluation of Quadriceps During Eccentric Decline Squat
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Sevim ACARÖZ CANDAN, Head of Department of Physiotherapy and Rehabilitation, Ordu University
Other Study IDs: OrduU6
Record Dates: First submitted 2019-12-06; First posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Patellar Tendinopathy
Keywords: eccentric squatting; electromyografic activation; exercise; patellar tendinopathy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies have generally investigated patellar tendon stiffness, cross-sectional area of patellar tendon, patellar tendon length, patellar force and patellafemoral forces during decline squat. However, there is just a few study about electromyographic (EMG) activity during the eccentric squating, which is about rectus femoris (RF) recruitment. In the present study the investigators primarly aimed to quantify the activation of RF, vastus lateralis (VL), and vastus medialis obliqus (VMO) during eccentric squat on different decline angle (0, 5°, 10°, 15°, 20°). An additional purpose of our study was to compare the changes in muscle activation at various arc of knee flexion motion (degrees of 0-30, 30-60, 60-90, 0-60, 30-90, 0-90).The investigators hypothesised that the recruitment of RF, VL, and VMO during eccentric squat would differ according to decline angle and arc of motion.

DETAILED DESCRIPTION:
The squat procedure in each condition will be repeated 10 times on a treadmill. The treadmill will be used to adjust the degree of decline in a standard manner. There will be a metronome to keep the speed of exercise in the same rhythm. All squats will be performed with a weighted barbell. The weight of it will be set as in ratio 30% of the participant's body weight

ELIGIBILITY:
Inclusion Criteria:

* had exercised regularly (>3 days in a week) for at least six months.
* older than 18 years old.

Exclusion Criteria:

* had patellofemoral pain, knee pain otherwise unrelated to the knee extensor mechanism and other injuries that would restrict performance of the tasks (e.g. ankle pathology).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asymptomathic older than 18 years, voluntary subjects who are students in a high school of physical education and sports.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-12-15 (Estimated); Primary Completion 2019-12-21 (Estimated); Study Completion 2019-12-22 (Estimated)

PRIMARY OUTCOMES:
Electromyographic measurement of muscle activation | 50 minutes
  Surface electromyographic (EMG) system (Noraxon Telemyo DTS System, Scottsdale, USA) will be use to measure the muscle activation ratios of RF, VL, and VMO. Electrodes will be placed according to Surface EMG for noninvasive assessment of muscles (SENIAM) recommendations on the dominant leg.
  The muscle activation during eccentric phase of the decline squat for RF, VL, and VMO will be determined. The decline squat will be performed under different conditions (various decline angle: 0, 5, 10,15, 20 degree) The muscle activation will also be investigated within various arc of motion of knee flexion (0-30, 30-60, 60-90, 0-60, 0-90, 30-90) which is determined using the motion analysis system (Noraxon, MYOmotion Scottsdale, USA).
Maximal voluntary isometric contractions (MVICs) | 5 minutes
  MVICs for the RF, VL, and VMO at their manual muscle test positions will be assessed within 3 trials, which lasts 5 seconds. The muscle test position will be standardized 90 degrees hip flexion and 60 degrees knee flexion. One minute a rest period will be between each trial. The peak EMG amplitude will be used for the normalization.
Normalized EMG values | 5 minutes
  The amount of muscle activation in each condition will be proportioned to MVICs value for normalization using a calculator. The value will be represented in percentile (%).

SECONDARY OUTCOMES:
Weight | 1 minute
  The participant's weight will be determined a weighing machine inkilogram.
Height | 1 minute
  The participant's height will be measured in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Acaröz Candan, PhD, Principal Investigator — Ordu University
Locations (1):
- Sevim ACARÖZ CANDAN, Ordu, Altinordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No